CLINICAL TRIAL: NCT06268704
Title: Particulate Versus Non-Particulate Corticosteroid in Sacroiliac Joint Injection: A Randomized Prospective Study
Brief Title: Particulate vs. Non-Particulate Steroid for Sacroiliac Joint Injection
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, rehsanian, Assistant Professor and Vice Chair of Clinical Research, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNM HRRC #23-503
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Sacroiliac Joint Dysfunction; Sacro-Iliac Spondylosis
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; Methylprednisolone; Methylprednisolone Hemisuccinate; Methylprednisolone Acetate; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Non-Particulate Steroid (Experimental): Patients in this arm will receive an injection of 1 milliliter of 2% lidocaine with 10 milligrams of dexamethasone to one or both sacroiliac joints. If participants initially achieve relief from the injection but then have a return of pain they may be offered a second injection with the same drug at the same dose.
  Interventions: Drug: Dexamethasone; Drug: 2% Lidocaine HCl Injection
- Particulate Steroid (Active Comparator): Patients in this arm will receive an injection of 1 milliliter of 2% lidocaine with 40 milligrams of methylprednisolone to one or both sacroiliac joints. If participants initially achieve relief from the injection but then have a return of pain they may be offered a second injection with the same drug at the same dose.
  Interventions: Drug: Methylprednisolone; Drug: 2% Lidocaine HCl Injection

INTERVENTIONS:
Drug: Dexamethasone — This is a non-particulate steroid commonly used to treat SI joint pain.
  Other Names: Ozurdex; Maxidex; DexPak
  Arms: Non-Particulate Steroid
Drug: Methylprednisolone — This is a particulate steroid commonly used to treat SI joint pain.
  Other Names: Solu-medrol; Depo-Medrol; Medrol
  Arms: Particulate Steroid
Drug: 2% Lidocaine HCl Injection — Lidocaine is a local anesthetic used in SI joint injection procedures to numb the procedure site and helps to confirm SI joint dysfunction when injected with the steroid medication into the SI joint.
  Other Names: Lignocaine; Xylocaine

SUMMARY:
This study will compare two different corticosteroids (dexamethasone and methylprednisolone) for use in sacroiliac joint injections to treat SI joint pain.

DETAILED DESCRIPTION:
Patients who are screened for inclusion will be randomized into one of two groups; dexamethasone or methylprednisolone. Patients will report their pain immediately after the procedure to confirm the diagnosis of sacroiliac joint pain, then be followed for three months to compare the efficacy and safety of the two medications.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18, capable of understanding and providing consent in English, capable of complying with the outcome instruments used, capable of attending all planned follow up visits
* Unilateral low back/buttocks pain of at least 2 weeks.
* Patient reported 7 day average of numeric pain rating score (NPRS) low back/buttocks pain of at least 5/10 at baseline evaluation
* Clinical diagnosis of sacroiliac joint pain as diagnosed by a board certified Physiatrist including history of low back/buttocks pain and at least 2 positive physical exam findings (including positive fortin finger sign, pain with palpation of posterior superior iliac spine, positive FABER's test, positive Gaenslan's test, positive sacral distraction, positive thigh thrust, positive lateral compression, positive sacral thrust)
* Patient consents to sacroiliac joint corticosteroid injection in a shared decision-making process with the treating physician.
* 80% or more relief of index pain within first 5-15 minutes after injection

Exclusion Criteria:

* Clinical suspicion of alternative process is greater than clinical suspicion of sacroiliac joint pain
* Those receiving remuneration for their pain treatment (e.g., disability, worker's compensation).
* Those involved in active litigation relevant to their pain.
* Those unable to read English and complete the assessment instruments.
* Those unable to attend follow up appointments
* The patient is incarcerated.
* History of prior sacroiliac joint fusion
* Progressive lower extremity neurologic deficit (from active radiculopathy, unhealed radiculopathy, or neuromuscular disease)
* Sacroiliac joint steroid injection within the prior 12 months
* 2 Positive lumbar medial branch blocks within the past 12 months
* Radiofrequency ablation of the lumbar spine within the past 12 months
* Lumbar facet steroid injections within the past 12 months
* Prior epidural steroid injection within the prior 3 months in any location within the spine.
* Possible pregnancy or other reason that precludes the use of fluoroscopy.
* Allergy to steroid, contrast media, or local anesthetics.
* BMI>40.
* Systemic inflammatory arthritis (e.g., rheumatoid arthritis, ankylosing spondylitis, lupus).
* Active infection or treatment of infection with antibiotics within the past 7 days.
* Medical conditions causing significant functional disability (e.g., stroke, decompensated ---COPD, decompensated heart failure)
* Chronic widespread pain or somatoform disorder (e.g. fibromyalgia).
* Addictive behavior, severe clinical depression, or psychotic features.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain using Numeric Pain Rating Score | 3 months
  Numeric pain rating score is an 11 point scale (0-10) filled out on a form indicating the degree to which the patient experiences pain to assess efficacy of the injection. In this scale a 0, the minimum score, indicates no pain at all with a 10, the maximum score, being the worst pain imaginable. In this study a 50% or greater reduction in numeric pain rating score is considered a successful outcome while failure to achieve at least a 50% improvement as compared to their numeric pain rating score prior to the procedure is considered a poor outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Reza Ehsanian, MD, PhD, Principal Investigator — University of New Mexico Department of Anesthesiology and Critical Care
Locations (1):
- University of New Mexico Hospital, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No